CLINICAL TRIAL: NCT03896113
Title: Influence of the Celecoxib Administration Before Surgery for Endometrial Cancer on Indoleamine 2,3-dioxygenase 1 (IDO1) Tumor Expression and Immune Cells Tumor's Infiltration
Brief Title: Neoadjuvant Celecoxib in Newly Diagnosed Patients With Endometrial Carcinoma
Acronym: CELEBRIDO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUC19-001
Record Dates: First submitted 2019-03-08; First posted 2019-03-29 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Endometrium Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Celecoxib; Cyclooxygenase 2

STUDY DESIGN:
Intervention Model Description: Open label, proof of concept phase II study. One arm, no placebo: All the patient will received the treatment and biopsies before and after the treatment will be compared regarding Indoleamine 2,3-dioxygenase 1 (IDO-1) expression and Immune T cells infiltration of the tumour
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Celecoxib (Experimental): Patients with confirmed primary endometrioid adenocarcinoma eligible for first line curative surgery will receive celecoxib 400 mg twice a day, for 15 days before the curative surgery for their endometrial cancer. The patients will undergo an endometrial biopsy at the inclusion and during the surgery.
  Interventions: Drug: Celecoxib 200mg capsule

INTERVENTIONS:
Drug: Celecoxib 200mg capsule — Patient confirmed with endometrial cancer will received twice daily 200 mg Celecoxib, 15 days before the surgery.
  Other Names: Cyclooxygenase-2 (COX-2) inhibitor

SUMMARY:
Indoleamine 2,3 dioxygenase 1 (IDO 1) is the major enzyme catabolising the Tryptophan outside the liver. It has been shown that its plays a important role in generating a immunosuppressive micro-environment in tumors. IDO expression has been shown by Hennequart et al. to be driven by Cyclooxygenase-2 (COX-2) expression. The investigator's team also shown that anti-COX2, celecoxib, can in a xenograft models of ovarian cancer decrease IDO1 expression and result in an infiltration of the tumor by T cells. The investigator proposed then to conduct a proof of concept study to evaluate the effect of pre-operative short administration of Celecoxib on IDO expression and Immune cells tumors infiltration, in patients with endometrial cancer. Indeed, this tumor type is well known to express frequently a high level of IDO.

DETAILED DESCRIPTION:
Indoleamine 2,3-dioxygenase 1 (IDO1) is an enzyme that regulates immune responses by degrading tryptophan, which is required for efficient T-cell activation. IDO1 expression is limited in normal tissues but is induced by IFN-gamma in inflammatory tissues, to prevent excessive T-cell activity. The investigator's collaborators previously reported that IDO1 is expressed in many human tumours, and that pharmacological inhibition of IDO1 leads to immune rejection of IDO1+ mouse tumours. Based on these results, IDO1 inhibitors are now in clinical development. A first inhibitor, Epacadostat, showed encouraging results combined with anti- Programmed Cell Death -1 (PD-1) antibodies. Tumoural expression of IDO1 can be induced by IFN-gamma, which is produced by tumour-infiltrating lymphocytes (TIL), and represents a mechanism of adaptive immune resistance. However, other tumours express IDO1 in the absence of TIL and Interferon-gamma (INF gamma). This seems to be particularly frequent in endometrial carcinoma. This constitutive IDO1 expression prevents T-cell infiltration and represents a mechanism of intrinsic immune resistance. The investigator's collaborators recently showed that constitutive tumoural expression of IDO1 was triggered by cyclooxygenase-2 (COX-2) and mediated by autocrine prostaglandin-E2 (PGE2) signaling via the Protein Kinase C (PKC) and phosphoinositide 3-kinase (PI3K) pathways. Constitutive IDO1 expression was reduced by COX-2 inhibitors in vitro. Celecoxib is a well-known and widely used anti-inflammatory drug. It is a specific inhibitor of COX-2. In vivo, celecoxib induced immune rejection of IDO1-expressing human tumour xenografts, while reducing IDO1 expression and promoting T-cell infiltration. These preclinical results suggest that COX-2 inhibition in patients carrying tumours expressing IDO1 constitutively will decrease IDO1 expression, increase T-cell infiltration and might increase responsiveness to anti-PD-1/ Programmed Cell Death Ligand-1(PD-L1) therapy and thereby exert enhanced anti-tumour activity. The investigators wish to obtain clinical evidence that celecoxib can induce these first two effects

ELIGIBILITY:
Key Inclusion Criteria:

* Women > 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2
* Adequate renal, hepatic and haematologic functions as defined by laboratory parameters.
* Agrees to undergo additional endometrial biopsies for scientific purposes.

Key Exclusion Criteria:

* Known hypersensitivity or intolerance to celecoxib
* Active, known or suspected autoimmune disease. Vitiligo, type I diabetes mellitus, residual hypothyroidism controlled by hormone substitution therapy, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are allowed.
* Positive hepatitis B or C, HIV, and pregnancy tests.
* Immunosuppressive treatment

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-11-13 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Reduction of tumoural cells expression IDO after celecoxib treatment. If more than 10% of all the tumoural cells have a staining for IDO, the tumour is considered as IDO (+), if less than 10%. | after 15 days of celecoxib administration
  Reduction of Tumoral IDO expression after Celecoxib treatment by immunohistochemistry, digital identification of the cells and phenotype and computer count of IDO positive cells inside de tumour (then total number compared before and after the treatment). If more than 10% of all the tumoural cells have a staining for IDO, the tumour is considered as IDO (+), if less than 10%, it is considered as (-).
  Based on animal models, the treatment with celecoxib should decreases IDO expression in tumoural cells, allowing an immune cells tumoural's infiltration.
Modification of tumoural T Cells infiltration after the treatment with celecoxib. The number of Cluster of Differenciation (CD) 4 and CD8 T cells will be counted before and after the treatment. | after 15 days of celecoxib administration
  Observed the modification of the T cell tumoral's infiltration after the celecoxib treatment by immunohistochemistry, digital identification of the cells and phenotype and computer count of the different T cells population inside de tumour (then total number compared before and after the treatment). The number of CD4 and CD8 T cells will be counted before and after the treatment and the median of all the sample before and after the treatment will be compared to assess if there is a significant difference of total number of T cells before and after the treatment. Unit= nombre of CD4 and CD8 T Cells. Based on animal model, the investigators expect to have a significant increase of T cells infiltration after the celecoxib treatment

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Event Version 4.0 (CTCAE v4.0). | from the first intake of the celecoxib to one day after the surgery
  Assessment and scaling of adverse events according to CTCAE v4.0, Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated;
  Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to Adverse Event.

CONTACTS AND LOCATIONS:
Overall Officials: Benoit van den Eynde, PhD, Study Director — Institut de Duve - UCL; Nicolas Van Baeren, PhD, Study Director — Institut de Duve- UCL; Jean-François Baurain, PhD, Study Chair — Cliniques universitaire St-Luc; Pierre van der Bruggen, PhD, Study Chair — Institut de Duve
Locations (2):
- Belgium (2):
  - Cliniques Universitaires Saint Luc, Brussels
  - Gasthuisberg - KULeuven, Leuven

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hennequart M, Pilotte L, Cane S, Hoffmann D, Stroobant V, Plaen E, Van den Eynde BJ. Constitutive IDO1 Expression in Human Tumors Is Driven by Cyclooxygenase-2 and Mediates Intrinsic Immune Resistance. Cancer Immunol Res. 2017 Aug;5(8):695-709. doi: 10.1158/2326-6066.CIR-16-0400. Epub 2017 Jul 21. PMID 28765120